CLINICAL TRIAL: NCT05884944
Title: Effects Of Osteopathic Manipulative Medicine(OMM) On Lower Extremity Muscle Characteristics In Parkinson's Disease(PD) Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Sheldon Yao, Chair, Professor OMM Department, New York Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BHS-1850
Record Dates: First submitted 2023-03-30; First posted 2023-06-01 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease; Osteopathy in Diseases Classified Elsewhere
Keywords: Osteopathic Manipulative Medicine
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group- OMM- Muscle energy (Experimental): For the OMM treatment group, an osteopathic manipulative treatment protocol will be applied to the lower extremities, specifically muscle energy technique (MET) to the hip, knee, and ankle bilaterally based on the protocol from Atlas of Osteopathic Techniques. The adductor, extensor, and flexor muscles of the hip joint will be treated, the extensors and flexors of the knee joint will be treated, and the plantar and dorsiflexion muscles of the ankle will be treated
  Interventions: Procedure: Experimental: Interventional Group- OMM- Muscle energy
- Control Group- Sham- Light touch, not reaching restrictive barrier (Sham Comparator): Joint articulation without engaging joint barriers The sham group will serve as the control group and will receive a sham-control procedure as outlined in the paper by Wells, et al in which they will undergo voluntary ROM and then passive movement with the same joint movements without reaching their barrier and no isometric contraction (Wells et al. 1999) The proposed sham procedure will occupy the same amount of time as MET treatment.
  Interventions: Procedure: Sham- Light touch, not reaching restrictive barrier

INTERVENTIONS:
Procedure: Sham- Light touch, not reaching restrictive barrier — Sham- Light touch, not reaching restrictive barrier For the control group, the subjects hip, knee, and ankle joints will be moved bilaterally 3 times into each plane to mimic the OMM muscle energy treatment. The joint will be moved in each plane of motion without reaching the joint barrier. The hip joint will be moved into adduction, extension, and flexion, the knee joint will be moved into extension and flexion, and the ankle will be moved into plantarflexion and dorsiflexion 3 times in each direction without reaching the barrier passively.
  Arms: Control Group- Sham- Light touch, not reaching restrictive barrier
Procedure: Experimental: Interventional Group- OMM- Muscle energy — The interventional group will received Osteopathic Manipulative Medicine, specifically Muscle energy treatment. An osteopathic manipulative treatment protocol will be applied to the lower extremity joints bilaterally. Muscle energy technique (MET) will be applied to the hip, knee, and ankle bilaterally based on the protocol from Atlas of Osteopathic Techniques. The adductor, extensor, and flexor muscles of the hip joint will be treated, the extensors and flexors of the knee joint will be treated, and the plantar and dorsiflexion muscles of the ankle will be treated. Muscle energy is a direct active treatment asking the subject to move their joint in a direction against a counterforce by the treatment provider for 3 times for 3 seconds and repeating the procedure 3 times and afterwards a passive stretch to the joint is applied by the provider.
  Arms: Interventional Group- OMM- Muscle energy

SUMMARY:
The purpose of the study is to investigate the effects that Osteopathic Manipulative Medicine has on lower extremity muscle characteristics in PD. Muscle stiffness, range of motion, and gait will be measured.

Participants will be asked to attend one in person session at the NYIT Academic Health Care Center. Participants will be randomly assigned to a control or experimental group. After a visit with the treating physician, both groups will have muscle stiffness tested using a myotonometry meter via a MyotonPRO device, gait measured while walking on a treadmill for 2 minutes before and after treatment, and range of motion tested using a goniometer. One week after the visit, participants will be asked to complete a brief survey over the phone with one of the study investigators.

DETAILED DESCRIPTION:
Parkinsonism, most commonly caused by Parkinson's disease (PD), is a syndrome characterized by rest tremor, rigidity, bradykinesia, and postural instability. Gait speed and endurance directly inhibit the independence and community engagement for those with Parkinson's disease (PD). Pain was ranked as one of the most troublesome nonmotor symptoms associated with PD. Rigidity is commonly associated with pain in patients with PD. Osteopathic medicine treats somatic dysfunction which is the impaired function of body components including the somatic, skeletal, myofascial, vascular, lymphatic, and neural systems. Osteopathic manipulative treatment (OMT) will be applied to the lower extremity (LE), specifically muscle energy technique (MET) to the hip, knee, and ankle bilaterally. A sham control group will receive passive range of motion (PROM) joint movement of the hip, knee, and ankles bilaterally without reaching joint physiologic barrier. Muscle and gait parameters, ROM, Timed Up & Go (TUG) and LE functionality will be assessed and juxtaposed. Based on preliminary results of muscle measurements, stiffness and relaxation improved in a patient with PD before and after LE OMT and demonstrated to be feasible. Investigators intend for the patients who receive OMT to improve LE muscle quality, gait, ROM, TUG, and daily functionality. Through this research Investigators hope to demonstrate that OMM as a supplemental treatment regimen can improve quality of life in those living with PD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease as per a neurologist, a severity of 2-4 on the Hoehn and Yahr (H-Y) Scale
* Able to receive OMM
* Able to be in a supine and prone position for MyotonPRO measurements
* Able to ambulate for gait measurements
* Have musculoskeletal complaints of leg pain/cramping or gait abnormalities due to their PD

Exclusion Criteria:

* Presence of severe fasciculations based on clinical judgment due to interference with measurements
* Gait disorders not attributed to PD
* Presence of other medical neurologic diagnoses that can affect outcome measures such as muscle tone/stiffness and ambulation (ie stroke, multiple sclerosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mechanical stress via the MyotonPro | Pre and Post intervention(1 hour)- change is being assessed
  Mechanical Stress Relaxation Time [ms]
Dynamic Stiffness via the MyotonPro | Pre and Post intervention(1 hour)- change is being assessed
  Dynamic Stiffness [N/m]
Step Cycle time via the Biodex Gait Trainer 3 | Pre and Post intervention(1 hour)- change is being assessed
  Gait will be investigated utilizing the Biodex Gait Trainer 3. Measurements will be taken during a two minute walk before and after treatment or sham protocol at the visit. Step cycle time- Cycles/ second
Average step length via the Biodex Gait Trainer 3 | Pre and Post intervention(1 hour)- change is being assessed
  Gait will be investigated utilizing the Biodex Gait Trainer 3. Measurements will be taken during a two minute walk before and after treatment or sham protocol at the visit.
  Average Step length in Cm
Step Symmetry- time on each foot via the Biodex Gait Trainer 3 | Pre and Post intervention(1 hour)- change is being assessed
  Gait will be investigated utilizing the Biodex Gait Trainer 3. Measurements will be taken during a two minute walk before and after treatment or sham protocol at the visit. Measurements include step symmetry via the time on each foot in percentage(%)
Goniometer- Hip ROM (Flexion and Extension) | Pre and Post intervention(1 hour)- change is being assessed
  A goniometer will be used to assess range of motion of the hip in degrees
Goniometer- Hip ROM Flexion | Pre and Post intervention(1 hour)- change is being assessed
  A goniometer will be used to assess range of motion of the hip in degrees
Goniometer- Hip ROM Extension | Pre and Post intervention(1 hour)- change is being assessed
  A goniometer will be used to assess range of motion of the hip in degrees
Goniometer- Knee ROM - Flexion | Pre and Post intervention(1 hour)- change is being assessed
  A goniometer will be used to assess range of motion of the Knee in degrees
Goniometer- Knee ROM - Extension | Pre and Post intervention(1 hour)- change is being assessed
  A goniometer will be used to assess range of motion of the knee in degrees
Goniometer- Ankle ROM- Dorsiflexion | Pre and Post intervention(1 hour)- change is being assessed
  A goniometer will be used to assess range of motion of the ankle in degrees
Goniometer- Ankle ROM- Plantarflexion | Pre and Post intervention(1 hour)- change is being assessed
  A goniometer will be used to assess range of motion of the ankle in degrees
The Timed Up & Go- 3 Meter walk | Pre and Post intervention(1 hour)- change is being assessed
  The Timed Up & Go (TUG) test measures one's ability to rise up from a seated chair position, walk 3 meters, turn, walk back, and sit down in the chair- measure in seconds

SECONDARY OUTCOMES:
Lower Extremity Functional Scale (LEFS) | Pre intervention and 1 week Post intervention - change is being assessed
  Lower Extremity Functional Scale (LEFS) will be used to assess difficulty with daily activities as a result of lower extremity dysfunction. Minimum value is 9 Maximum value is 80. The higher the score, the lower the disability.

CONTACTS AND LOCATIONS:
Locations (1):
- NYIT College of Osteopathic Medicine, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No